CLINICAL TRIAL: NCT06559813
Title: Step by Step - Pilot Study of Cognitive Behavior Therapy With Role-plays in Virtual Reality for Parents of Children With Anger, Oppositional or Aggressive Behaviors
Brief Title: Pilot Study of Parent Training With Role-plays in Virtual Reality for Parents of Children With Behavior Problems
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: PRIMA (Unknown); Psykologpartners (Unknown)
Responsible Party: Principal Investigator, Pia Enebrink, Associate professor, Karolinska Institutet
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-00813-01 - Parents
Record Dates: First submitted 2024-08-14; First posted 2024-08-19 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Child Behavior Problem; Disruptive Behavior; Oppositional Defiant Disorder; Conduct Problems; Aggression; Parent-Child Relations
Keywords: Disruptive Behavior; Child Behavior Problem; Parenting; Virtual Reality
MeSH Terms: conditions — Problem Behavior; Oppositional Defiant Disorder; Aggression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Parent training with cognitive behavior therapy and virtual reality (Experimental): A parent training program with between 6 and 10 individual, face-to-face, weekly sessions with parent
  Interventions: Behavioral: Step-by-step: A cognitive behavioral parent program with role-plays in virtual reality

INTERVENTIONS:
Behavioral: Step-by-step: A cognitive behavioral parent program with role-plays in virtual reality — A parent training program based on social learning theory and cognitive behavioral therapy (CBT), incorporating virtual reality for training in brief role plays. The program includes similar strategies as other common CBT-parent training programs for parents of children with behavior problems, with the difference that virtual reality is used as an additional way to practice skills.

SUMMARY:
The main aim of this pilot trial is to evaluate preliminary effects and feasibility of a new parent training program for parents of children aged 8-16 years with disruptive behavior (e.g., angry, aggressive or defiant behavior). The parent training program is based on cognitive behavioral therapy (CBT) and includes practicing of skills in virtual reality (VR).

The main questions the project aims to answer are:

* What are the preliminary effects of the CBT-VR parent training program?
* What is the level of parent engagement in the CBT-VR parent training program?
* What are the experiences of parents and therapists of the CBT-VR parent training program?

The CBT-VR parenting program is delivered at clinics during individual sessions. Parents will answer quantitative measurements before, during, and after treatment. Within-group analyses will be conducted to examine experiences and preliminary effects of the program. Parents and clinicians are also asked to participate in a qualitative interview after the program has ended.

DETAILED DESCRIPTION:
BACKGROUND:

Parent training programs based on cognitive behavioral therapy (CBT) have shown positive effects for reducing child behavior problems, such as oppositional defiant and aggressive behaviors, and are often recommended as a first intervention. The focus of CBT-based parenting programs are e.g. to reduce negative parent-child interactions and increase positive communication.

Recently, studies have evaluated CBT with the addition of exercises and role-playing in virtual reality (VR), for instance for adults with anxiety or anger. VR can provide a safe and gradual platform to practice in environments and situations. The present project evaluates a CBT-based parenting program, which includes practicing of skills in VR.

PURPOSE AND RESEARCH QUESTIONS:

The aim of this project is to evaluate preliminary effects and feasibility of a CBT-VR parent training program. The specific research questions are as follows:

1. What are the preliminary effect of the CBT-VR parent training program on children's behavioral problems, well-being, parents' emotion regulation, parenting strategies, and family conflicts?
2. What is the level of parent engagement in the CBT-VR parent training program (e.g., the number of sessions, exercises, homework completion and dropout rates)?
3. What are the experiences of parents and therapists of the CBT-VR parent training program (e.g., its effectiveness, acceptability, usefulness as well as relevance of the strategies taught)?

METHODS:

This project consists of a small pilot study of a CBT-VR parent training program for parents with children aged 8-16 years (n=10 families). The design is based on a mixed-methods approach. Evaluation of the intervention is conducted using within-group design (repeated measurements before, during, and after the intervention).

Parents will be recruited through clinics and advertisements. They are directed to a webpage with information about the study and contact information to the researchers. Parents give written informed consent to participate. When parents are interested in participating, a member of the research team will contact the participant for screening of inclusion and exclusion criteria. Clinicians at the respective clinics will be invited to answer questions regarding experiences of delivering the program.

The treatments are evaluated quantitatively by the parents using validated assessment forms/single questions before, during, and after interventions. Additionally, qualitative interviews will be conducted with parents and clinicians who provide consent to participating in an interview.

In another, separate study we evaluate CBT and role-plays in VR for children: "Pilot study of cognitive behavior therapy with role-plays in virtual reality for children with anger problems".

POWER CALCULATION:

The quantitative and qualitative data that will be collected with ten families is considered sufficient to provide understanding and preliminary insight into acceptability, usability, relevance, and effectiveness.

ANALYSES:

The plan is to compare changes during the intervention using paired t-tests, descriptive statistics, description of reliable and clinical change, and calculation of effect sizes. If appropriate, non-parametric alternatives will be employed. The qualitative analyses will be conducted using content analysis or thematic analysis.

ELIGIBILITY:
INCLUSION CRITERIA:

Parents:

* Parent of a child aged 8-16 years
* The parent perceives that the child has oppositional, angry or aggressive behaviors, and/or that there are parent-child conflicts at home.
* The child's behavior is elevated on a measure targeting behavioral problems (SDQ conduct problems subscale)

EXCLUSION CRITERIA

Parent treatment:

* Parent of a child under 8 years or over 16 years of age
* The child does not currently exhibit oppositional, angry or aggressive behaviors
* Child diagnosed with autism, serious depression, psychosis, eating disorder, or self-harm behaviors
* Parent has epilepsy or migraine

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Estimated)
Dates: Start 2024-08-19 (Estimated); Primary Completion 2024-11-25 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Parent: Mean change from baseline in behavior problems on parent-ratings of the Disruptive Behavior Disorder scale (oppositional defiant disorder subscale). | Pre- and post-intervention (10 weeks after the initiation of the intervention)
  The Disruptive Behavior Disorder subscale "Oppositional defiant disorder" is used for assessing children's behavioral problems. The subscale includes 8 items which are rated on a 4-point scale (0 to 3). The scale sum ranges från 0 to a total maximum sum of 24. A higher score indicates more behavior problems.
Parent: Mean change from baseline in parenting on parent-ratings of the Parenting Children and Adolescents Scale | Pre- and post-intervention (10 weeks after the initiation of the intervention)
  The Parenting Children and Adolescent Scale has three subscales: encouragement of positive behaviors, setting limits, proactive parenting behaviors. The 21 items are scored on a 5-point scale (1 to 5) and the total scale sum ranges from 21 to a maximum of 105, with a higher score indicating more positive parenting.
Parent: Mean change from baseline in parenting on parent-ratings of the Parenting Children and Adolescents Scale: Impact scale | Pre- and post-intervention (10 weeks after the initiation of the intervention)
  The 21 items included in the Parenting Children and Adolescents Scale each include a question of whether the item is experienced as a problem (yes/no). Total scale sum ranges between 0 and 21 with a higher sum indicating larger impact.

SECONDARY OUTCOMES:
Parent: Mean change from baseline in parent-ratings of child wellbeing on the KIDSCREEN-10 | Pre- and post-intervention (10 weeks after the initiation of the intervention)
  The KIDSCREEN-10 evaluates how parents perceive their child's/adolescent's health and well-being. The 10 items are scored on a 5-point scale (1 to 5). The total maximum sum ranges between 10 and 50 with a higher score indicating greater child wellbeing and health-related quality of life. The scale also includes an overall question about how the child is feeling in general.
Parent: Mean change from baseline in parent-ratings of child wellbeing on the Strengths and Difficulties Questionnaire (SDQ) | Pre- and post-intervention (10 weeks after the initiation of the intervention)
  The Strengths and Difficulties Questionnaire (SDQ) is used to assess mental health through a total difficulties score as well as through the five subscales (peer relationship problems, prosocial behavior, emotional symptoms, hyperactivity/inattention, conduct problems). The items are scored on a 3-point scale (0 to 2), and the total difficulties score is generated by summing all subscales except the prosocial scale. The summary score ranges from 0 to 40. Higher summary scores indicate more problems.
Parent: Mean change from baseline in parent-ratings of emotion regulation on the Difficulties in Emotion Regulation Scale-16 | Pre- and post-intervention (10 weeks after the initiation of the intervention)
  General emotion regulation ability will be measured with the Difficulties in Emotion Regulation Scale (brief version). The 16 items are scored on a 5-point scale (1 to 5), and the total summary score ranges between 16 and 80. A higher score indicates larger difficulties with emotion regulation.
Parent: Mean change from baseline in parent-ratings of parental emotion regulation on the Parent Emotion Regulation Scale | Pre- and post-intervention (10 weeks after the initiation of the intervention)
  Emotion regulation of the parent will be measured with the Parent Emotion Regulation Scale. The 20 items are scored on a 5-point scale (1 to 5). A total summary score ranges between 20 and 100 where a higher score indicates better regulation of emotions.
Parent: Mean change in parent-ratings of family warmth | Pre- and post-intervention (10 weeks after the initiation of the intervention)
  Family warmth is measured with 5 questions from the Family Check-Up Caregiver Assessment Scale. These are scored on a 5-point scale (1 to 5). Total maximum score ranges between 5 and 25. A higher score indicates a more positive relation.
Parent: Mean change in parent-ratings of family conflicts | Pre- and post-intervention (10 weeks after the initiation of the intervention)
  Family conflicts are measured with 3 questions from the Family Check-Up Caregiver Assessment Scale. These are scored on a 7-point scale (0 to 6). Total maximum score ranges between 0 and 18. A higher score indicates larger degree of conflicts.
Parent: Mean change in parent-ratings of parental satisfaction with the week | From baseline to post-intervention (during 6-10 weeks). Completed once a week at each session.
  Three questions scored 0 to 10 about parents' satisfaction with the week, with how they have been able to support their child and manage conflicts. Total maximum score ranges between 0-30, with a higher score indicating higher satisfaction.
Parent: Parental experiences of each session | From baseline to post-intervention (during 6-10 weeks). Completed once a week at each session.
  Four questions after each session about how the parent experienced the session and exercises. Rated on a scale 0-10, with a maximum total score ranging between 0 and 40. A higher score indicates greater satisfaction with the session.
Parent: Closing questions about the intervention | Post-intervention (measured 6 to 10 weeks after the initiation of the intervention)
  Closing questions to parents about satisfaction, relevance, and usefulness of the intervention. Parents respond to six questions rated on a scale 0-10, with a maximum total score ranging between 0 and 60. A higher score indicates greater satisfaction.
Use of the parent program: number of sessions, homework tasks, exercises | From pre- to post-intervention (10 weeks after the initiation of the intervention)
  A summary of the mean number of sessions, homework tasks and exercises completed during the program.
Use of the parent program: drop out rate | From pre- to post-intervention (10 weeks after the initiation of the intervention)
  The drop out from the program (number of participants).
Clinicians: Clinician perception of implementation | From pre- to post-intervention (during 6-10 weeks).
  Clinicians will respond to two questions rated 0-10 after each session about their implementation of the treatment session, higher scores indicating higher satisfaction (maximum weekly mean score is 20).
Parent, clinician: Experiences of the parenting program explored through separate, individual qualitative interviews with parent and clinician | Interviews are conducted after the program is completed, 10 weeks after the initiation of each program
  Qualitative interviews will explore parent's and clinician's experiences of the treatment. We will investigate satisfaction, feasibility, acceptability, and relevance of the program. The interviews with parents are partly based on an established scale, modified for this purpose, and self-constructed questions. Interviews with clinicians are based on self-constructed oral questions examining acceptability, relevance, feasibility and satisfaction.

OTHER OUTCOMES:
Background information | Pre-intervention
  Parents are asked for concise demographic information about themselves (e.g., age, education) and their child (e.g., age). A total of 8 questions.

CONTACTS AND LOCATIONS:
Overall Officials: Pia Enebrink, Principal Investigator — Karolinska Institutet